CLINICAL TRIAL: NCT04334304
Title: Evaluation of Standard and Robot Assisted Total Knee Arthroplasty with a Bicrucatie Retaining Prosthesis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient inclusion difficult.
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/1281 (BC-3831)
Record Dates: First submitted 2020-03-07; First posted 2020-04-06 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Osteo Arthritis Knee
Keywords: Total Knee Arthroplasty; Robot

STUDY DESIGN:
Intervention Model Description: Arm 1: Posterior Stabilized TKA without robot Arm 2: Posterior Stabilized TKA with robot Arm 3: Bicruciate retaining TKA without robot Arm 4: Bicruciate retaining TKA with robot
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Posterior Stabilized TKA without robot-assistance (Active Comparator): A TKA procedure will carried out: Posterior Stabilized TKA without robot-assistance
  Interventions: Procedure: Total Knee Prosthesis - type Posterior Stabilized
- Posterior Stabilized with robot-assistance (Experimental): A TKA procedure will carried out: Posterior Stabilized TKA with robot-assistance
  Interventions: Procedure: Robot-assisted Total Knee Arthroplasty; Procedure: Total Knee Prosthesis - type Posterior Stabilized
- Bicruciate retaining TKA without robot-assistance (Experimental): A TKA procedure will carried out: Bicruciate retaining TKA without robot-assistance
  Interventions: Procedure: Total Knee Prosthesis - type Bicruciate retaining
- Bicruciate retaining TKA with robot-assistance (Experimental): A TKA procedure will carried out: Bicruciate retaining TKA with robot-assistance
  Interventions: Procedure: Total Knee Prosthesis - type Bicruciate retaining; Procedure: Robot-assisted Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Total Knee Prosthesis - type Bicruciate retaining — A total knee arthroplasty will be performed with a bicruciate retaining implant (Journey II, XR). The control group will consist out of patients receiving a posterior stabilized implant (Journey II, BCS).
  Arms: Bicruciate retaining TKA with robot-assistance; Bicruciate retaining TKA without robot-assistance
Procedure: Robot-assisted Total Knee Arthroplasty — A total knee arthroplasty will be performed with robot-assistance (NAVIO).
  Arms: Bicruciate retaining TKA with robot-assistance; Posterior Stabilized with robot-assistance
Procedure: Total Knee Prosthesis - type Posterior Stabilized — A total knee arthroplasty will be performed with a bicruciate retaining implant (Journey II, XR). The control group will consist out of patients receiving a posterior stabilized implant (Journey II, BCS).
  Arms: Posterior Stabilized TKA without robot-assistance; Posterior Stabilized with robot-assistance

SUMMARY:
The first study goal is to compare the outcomes between Posterior Stabilized and Bicruciate Retaining TKA. Additionally, the second goal is to evaluate the effect of robot assisted surgery in both Posterior Stabilized and Bicruciate Retaining TKA.

ELIGIBILITY:
Inclusion Criteria:

* End stage osteoarthritis of the knee joint with failed conservative treatment

Exclusion Criteria:

* Previous ligament trauma
* Previous fracture of femur or tibia
* Fixed flexion contracture > 10°
* Flexion < 110°
* Coronal deformity > 15°
* Previous infection of the knee joint
* Ligament insufficiency
* Neurologic conditions

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Patient reported outcome measures | Preoperative
  The following patient reported outcome measures will be evaluated: Knee Injury and Osteoarthritis outcome score. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Patient reported outcome measures | Preoperative
  The following patient reported outcome measures will be evaluated: Knee Society Score. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Patient reported outcome measures | Preoperative
  The following patient reported outcome measures will be evaluated: EuroQoL. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Patient reported outcome measures | Preoperative
  The following patient reported outcome measures will be evaluated: Pain Catastrophizing Scale. The score is a percentage score from 0 to 52, 0 representing no problems and 52 representing extreme problems.
Change in patient reported outcome measures | Postoperatively at 6 weeks, 6 months, 1 year and 2 years.
  The change for the following patient reported outcome measures will be evaluated (compared to preoperatively): Forgotten Joint Score. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Change in patient reported outcome measures | Postoperatively at 6 weeks, 6 months, 1 year and 2 years.
  The change for the following patient reported outcome measures will be evaluated (compared to preoperatively): Knee Injury and Osteoarthritis outcome score. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Change in patient reported outcome measures | Postoperatively at 6 weeks, 6 months, 1 year and 2 years.
  The change for the following patient reported outcome measures will be evaluated (compared to preoperatively): Knee Society Score. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Change in patient reported outcome measures | Postoperatively at 6 weeks, 6 months, 1 year and 2 years.
  The change for the following patient reported outcome measures will be evaluated (compared to preoperatively): EuroQoL. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Change in patient reported outcome measures | Postoperatively at 6 weeks, 6 months, 1 year and 2 years.
  The change for the following patient reported outcome measures will be evaluated (compared to preoperatively): Pain Catastrophizing Scale. The score is a percentage score from 0 to 52, 0 representing no problems and 100 representing extreme problems.

SECONDARY OUTCOMES:
Alignment | Preoperative and postoperatively at 6 weeks and 6 months.
  Coronal alignment on xrays. The lateral distal femoral angle (LDFA) will be evaluated. This is the angle between the mechanical femoral axis and the line between the distal articular surface of the femur. Additionally the medial proximal tibial angle (MPTA) will be evaluated. This is the line between the condylar surface and the mechanical axis of the tibia on a coronal radiograph.
Knee laxity | Preoperative and postoperatively at 1 year.
  Coronal knee laxity will be evaluated with stress examination. Coronal stress will be evaluated with a stress radiograph. The deviation between the neutral position and position under stress will be measured on a coronal radiograph. The angle between the joint lines will be measured on the coronal radiograph.
Knee laxity | Preoperative and postoperatively at 1 year.
  Sagittal knee laxity will be evaluated with stress examination. Sagittal knee laxity will be measured with an AP laxitymeter (GENOUROB; CE Marked). With a standardized setup, anteroposterior laxity can be obtained by measuring the anteroposterior deviation from the neutral position with up to 300N of force.
Knee kinematics in 3D after squat, knee flexion/extension, stair ascend and descend. | Postoperatively at 1 year.
  Knee kinematics in 3D obtained with fluoroscopy. Patients will be asked to perform squats, a flexion/extension movement, ascend and descend stairs. 3D motion of the prosthesis components can be obtained by projecting the 3D file of the prosthesis components onto the fluoroscopy images.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Victor, PhD, Study Chair — UZ Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No